CLINICAL TRIAL: NCT01571505
Title: Exploration of the Biologic Basis for Underperformance of Oral Polio and Rotavirus Vaccines in INDIA
Brief Title: Exploration of the Biologic Basis for Underperformance of Oral Polio and Rotavirus Vaccines in INDIA (PROVIDE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); National Institute of Cholera and Enteric Diseases, India (Other); University of Virginia (Other); University of Vermont (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: POLIO ROTA-02
Record Dates: First submitted 2012-03-28; First posted 2012-04-05 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Poliomyelitis; Tropical Enteropathy
Keywords: Oral vaccines; Vaccine Responsiveness; Tropical Enteropathy
MeSH Terms: conditions — Poliomyelitis; Sprue, Tropical | interventions — Aging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPV vaccination (Experimental): Randomized IPV vaccination to children at the age of 39 weeks.
  Interventions: Biological: IPV vaccination
- OPV vaccination (Placebo Comparator): Randomized OPV vaccination to children at the age of 39 weeks.
  Interventions: Biological: IPV vaccination

INTERVENTIONS:
Biological: IPV vaccination — Randomized IPV or OPV to children aged at 39weeks.
  Other Names: Rotavirus vaccination to children at 10 and 17 weeks of age.

SUMMARY:
Oral polio and rotavirus vaccines are significantly less effective in children living in the developing world. Tropical enteropathy, which is associated with intestinal inflammation, decreased absorption and increased permeability, may contribute substantially to oral vaccine failure in developing country settings. Other possible causes of oral vaccine underperformance include malnutrition, interference with maternal or breast milk antibodies, changes in gut microbiota, and genetic susceptibility.The primary Objective of this study is to determine whether decreased vaccine responsiveness to oral poliovirus or rotavirus vaccines is associated with the presence of tropical enteropathy.

DETAILED DESCRIPTION:
Intervention of this study is to vaccinate oral poliovirus vaccine and oral rotavirus vaccine to the child with two group; with inactivated poliovirus vaccine and without inactivated poliovirus vaccine. Rotavirus vaccines give to the child at 10 weeks of age and 17 weeks of age.

ELIGIBILITY:
Inclusion Criteria:

1. Mother willing to sign informed consent form.
2. Infant aged 0 to 49 days old.
3. No obvious congenital abnormalities or birth defects.

Exclusion Criteria:

1. Parents are not willing to have child's blood drawn.
2. Parents are planning to enroll child into another clinical study during the time period of this trial.
3. Mother not willing to have blood drawn and breast milk extracted.
4. Parents not willing to have field research assistant in home.
5. History of seizures or other apparent neurologic disorders.
6. Infant does not have proof of BCG and OPV since birth by immunization card.
7. History of acute illness and/or immunocompromised state of the child.
8. Immunocompromised or chronically ill mother

Ages: 42 Days to 49 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 372 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Vaccine immunogenicity of oral vaccines (Oral Polio Vaccine and Rotavirus Vaccine) with the presence of tropical enteropathy using Lactose/Mannitol ratio in urine. | Birth to one year
  Responsiveness of oral vaccines compare with Tropical Enteropathy and without Tropical Enteropathy; using lactose/mannitol ratio.

SECONDARY OUTCOMES:
Systemic immune responses (neutralizing antibodies) of impact of an inactivated polio vaccine (IPV) and polio vaccine boost following vaccination with oral polio vaccine (OPV). | Birth to one year
Mucosal immune responses (shedding OPV vaccine virus) of impact of an inactivated polio vaccine (IPV) and polio vaccine boost following vaccination with oral polio vaccine (OPV). | Birth to one year

CONTACTS AND LOCATIONS:
Overall Officials: Ayan Dey, Ph.D, Principal Investigator — International Vaccine Institute; William Petri, M.D, Principal Investigator — University of Virginia; Beth Kirkpatrick, M.D., Principal Investigator — University of Vermont; Suman Kanungo, M.D., Principal Investigator — National Institute of Cholera and Enteric Diseases, India; Ranjan K Nandy, M.D., Principal Investigator — National Institute of Cholera and Enteric Diseases, India
Locations (1):
- National Institute of Cholera and Enteric Diseases, Kolkata, India

REFERENCES:
- [Result] Kanungo S, Kim DR, Haldar B, Snider C, Nalavade U, Kim SA, Park JY, Sinha A, Mallick AH, Manna B, Sur D, Nandy RK, Deshpande JM, Czerkinsky C, Wierzba TF, Petri WA Jr, Ali M, Dey A. Comparison of IPV to tOPV week 39 boost of primary OPV vaccination in Indian infants: an open labelled randomized controlled trial. Heliyon. 2017 Jan 9;3(1):e00223. doi: 10.1016/j.heliyon.2016.e00223. eCollection 2017 Jan. PMID 28194449